CLINICAL TRIAL: NCT05096845
Title: A Global, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Phase III Clinical Study to Evaluate the Efficacy, Safety, and Immunogenicity of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) in Adults Aged 18 Years and Older
Brief Title: Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) Phase III
Acronym: COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TG2101V01
Record Dates: First submitted 2021-10-21; First posted 2021-10-27 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pandemic
Keywords: V-01
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V-01 COVID-19 Vaccine (Experimental): Intramuscular injection into the lateral deltoid of the upper arm Two doses, one each on Day 0 and 21 (+7 days), respectively.
  Interventions: Biological: Recombinant SARS-CoV-2 fusion protein vaccine (V-01)
- Placebo control (Placebo Comparator): Intramuscular injection into the lateral deltoid of the upper arm Two doses, one each on Day 0 and 21 (+7 days), respectively.
  Interventions: Other: Blank Preparation of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01)

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 fusion protein vaccine (V-01) — Appearance: creamy white suspension Dosage form: Suspension for injection Strength: 10 μg (0.5mL) /vial Vaccination route: intramuscular injection into the lateral deltoid of the upper arm Vaccination dosage: 10 μg Immunization schedule: two doses, one each on Day 0 and 21 (+7 days), respectively.
  Storage condition: store at 2~8°C protected from light Expiry date: 24 months after production date
  Other Names: V-01
  Arms: V-01 COVID-19 Vaccine
Other: Blank Preparation of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) — The dosage, appearance, administration method, and other aspects are consistent with that of investigational vaccine, except that no vaccine antigen is contained.
  Arms: Placebo control

SUMMARY:
A Global, Multi-center, Randomized, Double-Blind, Placebo-Controlled, Phase III Clinical Study to Evaluate the Efficacy, Safety, and Immunogenicity of Recombinant SARS-CoV-2 Fusion Protein Vaccine (V-01) in Adults Aged 18 Years and Older

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, placebo-controlled, parallel-group phase III clinical study. Approximately 22,500 participants aged 18 years and older will be enrolled in this study to evaluate the efficacy, safety and immunogenicity of recombinant SARS-CoV-2 fusion protein vaccine (code: V-01, hereinafter referred to as V-01).

The eligible participants will be randomized in a 2:1 ratio into investigational vaccine group (V-01) and placebo group, with random stratification factors including 1) age (18-59 years vs ≥60 years); 2) gender (male vs female); and 3) whether or not being enrolled into immunogenicity subgroup (yes vs no). The participants will receive investigational vaccine V-01 or placebo on two doses schedule (one dose each on day 0 and 21, with +7 days' time window for the second dose).

ELIGIBILITY:
Inclusion Criteria:

The participants can be enrolled only all of the following criteria are met:

1. Voluntarily participate in this study and sign the informed consent form;
2. Adults aged 18 years and older, male or female;
3. According to the assessment of the investigator, the participant has a stable medical condition (which is defined as no significant changes in therapy or hospitalization caused by disease aggravation within 3 months before enrollment) and is able to and willing to follow the requirements of the protocol.
4. Males of reproductive potential and females of child-bearing potential voluntarily agree to take effective and acceptable contraceptive methods from the signing of informed consent form to 12 months after full-course immunization; females of child-bearing potential have a negative pregnancy test at screening and at the day of vaccination.

Exclusion Criteria:

Participants meeting any of the following exclusion criteria will not be allowed to participate in this study:

1.History of previous COVID-19 infection; 2.Positive result for RT-PCR test in the screening period or specific antibody IgG or IgM meet the following criteria:

1. If IgG is positive, the participant will be excluded regardless of the results of other indexes.
2. If IgG is negative and IgM is positive, it will be determined whether or not to enroll such participant after the result of RT-PCR test is obtained;
3. If both IgG and IgM are negative, the participant can be vaccinated without waiting for the RT-PCR test results.

3.History of severe acute respiratory syndrome (SARS), middle east respiratory syndrome (MERS), and other human coronavirus infections or diseases; 4.History of severe allergy to any vaccine, e.g., acute allergic reactions, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain etc., or be allergic to any components of V-01; 5.Any confirmed or suspected immunosuppression or immunodeficiency condition known from medical history, including human immunodeficiency virus (HIV) infection, asplenia; 6.Serious or uncontrolled cardiovascular diseases, nervous system disorders (e.g., Guillain-Barre syndrome), blood and lymphatic system disorders, immune system disorders, hepatorenal disorders, respiratory system disorders (e.g., active tuberculosis, pulmonary fibrosis), metabolic and skeletal systems disorders or malignant tumors (except for skin basal cell carcinoma or in situ carcinoma of uterine cervix that has been cured for more than 5 years); 7.Hereditary hemorrhagic tendency or coagulation dysfunction, or a history of thrombosis or hemorrhagic disease, or requirement of continuous use of anticoagulants; 8.Prior use of any medications to prevent COVID-19, e.g., use of antipyretics without pyrexia and any other symptoms; 9.A history of vaccination against SARS-CoV-2 (marketed or investigational); 10.Received attenuated live vaccine within 28 days before the first vaccination or any other vaccines (licensed or investigational) within 14 days before the first vaccination; 11.Injection of immunoglobulin and/or other blood products within 3 months before the administration of study vaccine; 12.Long-term use (continuous use >14 days) of glucocorticoids (≥10mg/day of prednisone or its equivalent dose) or other immunosuppressive agents; however, enrollment is allowed for the following conditions: inhaled or topical use of topical steroids, or short-term use (treatment course ≤14 days) of oral steroids; 13.Pregnant or breastfeeding women; 14.Planning to donate blood during the study period; 15.Suspected or known alcohol or drug dependence; 16.History of severe psychiatric disorders which may affect study participation; 17.Planning to permanently move from the local area before study completion or leave the local area for a long time during the period of study visits, so that the scheduled visits cannot be followed; 18.Those considered by the investigator as inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22500 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2023-06-14 (Estimated)

PRIMARY OUTCOMES:
The efficacy of V-01 for the prevention of symptomatic RT-PCR-positive COVID-19 (mild or above in severity) | More than 14 days (≥15 days) after full course immunization
  To evaluate the efficacy of the recombinant SARS-CoV-2 fusion protein vaccine (V-01) for the prevention of symptomatic RT-PCR-positive COVID-19 (mild or above severity) starting from at least 14 days (≥15 days) after full-course immunization (completing all vaccinations);
The incidence of adverse events (AEs) of V-01 | From the first vaccination to 28 days after full-course immunization
  To evaluate the incidence of adverse events (AEs) of recombinant SARS-CoV-2 fusion protein vaccine (V-01) from the first vaccination to 28 days after full-course immunization

SECONDARY OUTCOMES:
The efficacy of V-01 for the prevention of COVID-19 of severe or above in severity | More than 14 days (≥15 days) after full-course immunization;
  To evaluate the efficacy of the recombinant SARS-CoV-2 fusion protein vaccine (V-01) for the prevention of COVID-19 of severe or above severity starting from at least 14 days (≥15 days) after full-course immunization;
The efficacy of V-01 for the prevention of symptomatic RT-PCR-positive COVID-19 (mild or above in severity) | More than 14 days (≥15 days) after full-course immunization;
  To evaluate the efficacy of the recombinant SARS-CoV-2 fusion protein vaccine (V-01) for the prevention of symptomatic RT-PCR-positive COVID-19 (mild or above in severity) starting from more than 14 days after the first vaccination;
The efficacy of V-01 for the prevention of symptomatic RT-PCR-positive COVID-19 (mild or above in severity) in different age groups | More than 14 days (≥15 days) after full-course immunization;
  To evaluate the efficacy of the recombinant SARS-CoV-2 fusion protein vaccine (V-01) for the prevention of symptomatic RT-PCR-positive COVID-19 (mild or above in severity) starting from more than 14 days after full-course immunization in different age groups
The morbidity of suspected but not confirmed COVID-19 (negative or not detected) | More than 14 days (≥15 days) after full-course immunization;
  To evaluate the morbidity of suspected but not confirmed COVID-19 (negative or not detected)
The mortality caused by COVID-19 | More than 14 days (≥15 days) after full-course immunization;
  To evaluate the mortality caused by COVID-19
The hospitalization rate caused by COVID-19 | More than 14 days (≥15 days) after full-course immunization;
  To evaluate the hospitalization rate caused by COVID-19
The incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs) | From the first dose of recombinant SARS-CoV-2 fusion protein vaccine (V-01) to 12 months after full-course immunization
  To evaluate the incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs) occurred from the first dose of recombinant SARS-CoV-2 fusion protein vaccine (V-01) to 12 months after full-course immunization
The seroconversion rate of serum SARS-CoV-2 RBD protein-binding antibody, geometric mean titer (GMT) and geometric mean increase (GMI) | At day 28, month 3, month 6, and month 12 after full-course immunization
  1. To evaluate the seroconversion rate of serum SARS-CoV-2 RBD protein-binding antibody, geometric mean titer (GMT) and geometric mean increase (GMI) at day 28, month 3, month 6, and month 12 after full-course immunization (enzyme-linked immunosorbent assay [ELISA]);
  2. To evaluate the seroconversion rate of serum anti-SARS-CoV-2 neutralizing antibody, GMT and GMI at day 28, month 3, month 6, and month 12 after full-course immunization (live virus neutralization assay);

OTHER OUTCOMES:
The severity of COVID-19, so as to evaluate the vaccine-mediated antibody-dependent enhancement (ADE) | From the first dose of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-course immunization
  To evaluate the severity of COVID-19 of participants in the vaccine group versus the control group, so as to evaluate the vaccine-mediated antibody-dependent enhancement (ADE)
The correlation of immunogenicity and efficacy through evaluating the titer level of RBD protein-binding antibody in confirmed COVID-19 cases | From the first dose of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-course immunization
  To explore the correlation of immunogenicity and efficacy through evaluating the titer level of RBD protein-binding antibody in confirmed COVID-19 cases.
SARS-CoV-2 nucleic acid sequence in symptomatic and RT-PCR-positive COVID-19 cases | From the first dose of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-course immunization
  Genotypic analyses of SARS-CoV-2 nucleic acid sequence in symptomatic and RT-PCR-positive COVID-19 cases.
The immunogenicity of V-01 against new SARS-CoV-2 variants | From the first dose of recombinant SARS-CoV-2fusion protein vaccine (V-01) to 12 months after full-course immunization
  To explore the immunogenicity of V-01 against new SARS-CoV-2 variants

CONTACTS AND LOCATIONS:
Locations (25):
- Indonesia (4):
  - Andalas University Hospital, Padang
  - Medical Faculty of Mulawarman University, Samarinda
  - Medical Faculty of Padjadjaran University, Sumedang
  - Medical Faculty of UIN Syarif Hidayatullah, Tangerang
- Philippines (9):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - The Medical City- Iloilo, Iloilo City, Iloilo
  - Makati Medical Center, Makati City
  - University of the Philippines - Philippine General Hospital, Manila
  - East Avenue Medical Center, Manila
  - Lung Center of the Philippines, Manila
  - Mary Chiles General Hospital, Manila
  - Far Eastern University-Nicanor Reyes Medical Foundation Medical Center, Quezon City
  - St. Luke's Medical Foundation Medical Center, Quezon City
- Russia (12):
  - Central Clinical Hospital of the Russian Academy of Sciences, Engel's
  - Oris LLC, Moscow
  - Zvezdnaya Clinic, Moscow
  - UZI-4D Clinic LLC, Pyatigorsk
  - Institute of Medical Research LLC, Saint Petersburg
  - Lab. of molecular virology Smorodintsev Research Institute of Influenza MoH, Saint Petersburg
  - LLC "Uromed", Saint Petersburg
  - Medical Technologies, Saint Petersburg
  - N.P. Bechtereva Institute of the Human Brain of the Russian Academy of Sciences, Saint Petersburg
  - Research Center ECO Safety LLC, Saint Petersburg
  - State Budgetary Healthcare Institution "Nikolaevskaya hospital", Saint Petersburg
  - Strategic Medical Systems LLC, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided